CLINICAL TRIAL: NCT07122401
Title: A Multicenter, Randomized, Double-blind, Double-dummy, Phase III Study to Evaluate the Efficacy and Safety of MT1013 Versus Cinacalcet as Active Control in Secondary Hyperparathyroidism Patients on Maintenance Dialysis
Brief Title: Study of MT1013 for the Treatment of Patients With Secondary Hyperparathyroidism
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shaanxi Micot Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MT1013-III-C01
Record Dates: First submitted 2025-08-01; First posted 2025-08-14 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Secondary Hyperparathyroidism, Chronic Kidney Disease
MeSH Terms: conditions — Hyperparathyroidism, Secondary; Renal Insufficiency, Chronic | interventions — Cinacalcet

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MT1013 (Experimental): MT1013 is administered intravenously (IV) for 26 weeks; Dummy cinacalcet will be administered orally for 26 weeks.
  Interventions: Drug: MT1013
- Cinacalcet (Active Comparator): Cinacalcet is administered orally for 26 weeks. Dummy MT1013 is administered intravenously (IV) for 26 weeks.
  Interventions: Drug: Cinacalcet

INTERVENTIONS:
Drug: MT1013 — MT1013 + dummy cinacalcet
  Arms: MT1013
Drug: Cinacalcet — Cinacalcet + dummy MT1013
  Arms: Cinacalcet

SUMMARY:
MT1013 is a first-in-class dual-target agonist. This study is a multicenter, randomized, double-blind, double-dummy phase III clinical study being conducetd to evaluate the efficacy and safety of MT1013 compared with active control cinacalcet in secondary hyperparathyroidism patients on maintenance dialysis. Subjects will be 1:1 randomized to receive MT1013 or cinacalcet for 26 weeks. Evaluations of iPTH, Ca, P, BMD, and biomarkers will be done across the study period, to compare efficacy and safety of MT1013 to cinacalcet.

ELIGIBILITY:
Inclusion Criteria:

1. Participants capable of understanding written information ,willing to participate in, and provide a written informed consent;
2. Male or female, at least 18 years old, 18 kg/m^2 ≤BMI≤35 kg/m^2;
3. Receiving regular maintenance dialysis 3 times a week for at least 12 weeks prior to screening；
4. Dialysate calcium concentration≥1.25 mmol/L (2.5 mEq/L);
5. Subjects must have a confirmed diagnosis of Secondary Hyperparathyroidism (SHPT), with a mean pre-dialysis serum intact parathyroid hormone (iPTH) level ≥ 400 pg/mL (42.4 pmol/L), based on measurements from two non-consecutive days before dialysis, within 14 days prior to randomization;
6. Within 14 days prior to randomization, subjects must have serum calcium levels (measured pre-dialysis, or corrected serum calcium if albumin <40 g/L) ≥ 8.4 mg/dL (2.1 mmol/L) on two non-consecutive pre-dialysis measurements.

Exclusion Criteria:

1. Underwent parathyroidectomy within 6 months prior to screening, or anticipated parathyroidectomy, ablation or radiation during the study;
2. Gastrointestinal bleeding or peptic ulcer medical history within 6 months prior to screening;
3. New York Heart Association (NYHA) Class III or IV heart failure within 3 months prior to screening; Symptomatic arrhythmia within 6 months prior to screening; History of torsades de pointes (TdP).
4. QTcF interval >470 ms in males or >480 ms in females on screening ECG, or other clinically significant ECG abnormalities as determined by the Investigator (e.g., third-degree atrioventricular block, sick sinus syndrome, multifocal frequent ventricular premature contractions, ventricular tachycardia, atrial fibrillation, etc.).
5. Subjects with severe uncontrolled hypertension during the screening period are excluded, defined as systolic blood pressure >180 mmHg and/or diastolic blood pressure >110 mmHg despite optimal medical therapy prior to enrollment (excluding transient blood pressure abnormalities during dialysis).
6. History of seizure within 1 year prior to screening, or currently receiving treatment for seizure disorders;
7. Received oral cinacalcet or ivocalcet within 14 days prior to screening, or received Etelcalcetide injection treatment within 4 months prior to screening;
8. Any other condition that, in the Investigator's judgment, would make the subject unsuitable for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 424 (Estimated)
Dates: Start 2025-09-30 (Actual); Primary Completion 2026-11-26 (Estimated); Study Completion 2026-11-26 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with > 50% reduction from baseline in mean intact parathyroid (iPTH) | EAP（Week 22-27）
Percentage of participants with > 30% reduction from baseline in mean iPTH | EAP（Week 22-27）

SECONDARY OUTCOMES:
Change From Baseline in Bone Mineral Density | Week 27
Change from baseline in serum calcium | EAP（Week 22-27）
Change From Baseline in serum phosphorus | EAP（Week 22-27）
Safety and Tolerance | Up to Week 30
  Incidence and severity of TEAE/TESAE

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Shanghai, Shanghai Municipality, China